CLINICAL TRIAL: NCT05560360
Title: Study of the Pharmacokinetic Effects of Efavirenz on the Pharmacokinetics of SHR1459 in Healthy Subjects
Brief Title: A Trial of DDI Between SHR1459 and Efavirenz With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1459-I-110
Record Dates: First submitted 2022-09-27; First posted 2022-09-29 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: B-cell Tumors
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: Compare the pharmacokinetic effects of efavirenz on SHR1459 in healthy subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental)
  Interventions: Drug: SHR1459 tablet; Drug: Efavirenz tablet

INTERVENTIONS:
Drug: SHR1459 tablet — 100 mg/tablet; administered orally
Drug: Efavirenz tablet — 600 mg/tablet; administered orally

SUMMARY:
This study used a single-dose, open and fixed sequence design to compare the pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent before the test, and fully understood the test content, process and possible adverse reactions;
2. Age 18-45 (including threshold), male and female(at least 5 female subjects);
3. Weight ≥ 50 kg for male, weight ≥ 45 kg for female, body mass index (BMI): 18.5~30 kg/m2 (including critical value);
4. Heart rate 60-100 bpm;
5. Be able to communicate well with the investigators and understand and comply with the requirements in this study.

Exclusion Criteria:

1. Physical examination, vital signs, blood-routine examination, blood biochemistry, infectious disease screening, coagulation function, urine-routine examination, chest x-ray, B ultrasound and other examination results are abnormal and judged by the research doctor as clinically significant;
2. Glomerular filtration rate (GFR) < 90 mL/min/1.73 m2;
3. 12-lead ECG abnormalities, in which QTcF≥ 430 ms for men and QTcF≥ 450 ms for women, (the QTc interval is corrected by the Fridericia formula (QTcF = QT/(RR^0.33), RR is the standardized heart rate value, divided by heart rate of 60), sinus arrhythmias, sinus bradycardia, or other abnormalities are judged to be clinically significant by research physicians;
4. Those who have previously suffered from severe heart, lung, liver, kidney, blood, gastrointestinal, endocrine, immune, skin, neurological or psychiatric diseases or existing above diseases, which are judged by the research doctor to be unfit for participants;
5. Those who have undergone any surgery within 6 months prior to screening; or have previously undergone any surgery that affects the absorption of the drug in the stomach and intestines (including gastrectomy, bowel resection, gastric contraction surgery, etc.) and any surgery that affects liver function (including cholecystectomy, etc.);
6. Screening for any acute illness that has occurred within the month prior to the study as clinically significant;
7. Those with a specific history of allergies (e.g., asthma, urticaria, eczema, etc.), or have allergic constitution (those who are allergic to two or more drugs, foods, or environmental substances such as alcohol, milk, pollen, etc.), or those with a known history of allergies to SHR1459, efavirenz, or their excipients (SHR1459, see Appendix 2 for efavirenz excipients);
8. Have used any drugs that effect enzyme activity (e.g., antivirals, antifungals, antiplatelet aggregations, etc.) in the month prior to taking the study drug;
9. Have any prescription drugs, nonprescription drugs, vitamins, health supplements, proprietary Chinese medicines and herbs within month before taking the research drugs;
10. Persons with history of drug abuse/dependence in the past five years; Those with history of drug abuse or positive drug screening (including morphine, methamphetamine( methamphetamine), ketamine, ecstasy (methylenedioxyamphetamine), cocaine, cannabis (tetrahydrocannabinol acid) positive);
11. Alcohol abuse in the 3 months prior to screening, with an average daily intake of more than 15g of alcohol (equivalent to 145 mL of wine, 450 mL of beer or 43 mL of liquor with an alcohol content of 40%), and those who cannot abstain from alcohol during the trial, or those who have a positive alcohol breath screening;
12. Those who smoke more 5 cigarettes per day in the 3 months before screening or those who do not agree to quit smoking during the test, or those who are positive for urine nicotinic screen;
13. Those who donate blood or other reasons of bleeding cause the total loss of blood more than 200mL or receive blood transfusions within 3 months before screening;
14. Those who have used other experimental drugs or medical devices within 3 months before screening or who have used experimental biological macromolecules within 1 year;
15. From 48 hours before taking the study drug to the end of the study, subjects have xanthine-rich beverages (chocolate, coffee, tea, etc.) or food (animal liver, etc.), or grapefruit, star fruit and other fruits or juices that may affect metabolism;
16. Can not comply with the unified dietary arrangement or have special requirements for diet (such as intolerance to standard meal food, etc.); Or those who have strenuous exercise or are unwilling to accept the lifestyle required by the program; Or have other factors that affect the absorption, distribution, metabolism, excretion and other factors of the drug;
17. Those who have been vaccinated against the COVID-19 within one month before the first administration, or those who have received other vaccinations in the previous 3 months of screening;
18. Who have blood phobia and faint with acupuncture ; or those with poor vascular conditions, inability to embed needles or inability to tolerate venipuncture;
19. Lactating women, or female subjects who used long-acting estrogen or progestin injections (containing progestin-type intrauterine devices) or implant within 6 months prior to screening;
20. Women of childbearing potential (WOCBP) who have a positive serum pregnancy test;
21. Screening of persons who have had unprotected sex with their partners/sexual partners within one month prior to the screening;
22. Women of childbearing potential and sexual partners who have a WOCBP have a pregnancy plan or sperm donation, ovum donation program, or do not use medically approved contraception from the beginning of signing the informed consent form to 12 weeks after the last drug use;
23. Subjects who are judged by researchers to be unsuitable for participating in this test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of SHR1459: Cmax | Based on pre-dose, 0-24 hours post-dose sampling times
Pharmacokinetics parameters of SHR1459: AUC0-t | Based on pre-dose, 0-24 hours post-dose sampling times
Pharmacokinetics parameters of SHR1459: AUC0-inf | Based on pre-dose, 0-24 hours post-dose sampling times

SECONDARY OUTCOMES:
Pharmacokinetics parameters of SHR1459: Tmax | Based on pre-dose, 0-24 hours post-dose sampling times
Pharmacokinetics parameters of SHR1459: T1/2 | Based on pre-dose, 0-24 hours post-dose sampling times
Pharmacokinetics parameters of SHR1459: CL/F | Based on pre-dose, 0-24 hours post-dose sampling times
Pharmacokinetics parameters of SHR1459: Vz/F | Based on pre-dose, 0-24 hours post-dose sampling times
Incidence and severity of adverse events/serious adverse events (base on CTC AE 5.0) | Based on pre-dose to Day 24

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Lianyungang, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided